CLINICAL TRIAL: NCT05022303
Title: A Phase 2a (Proof of Concept), Randomized, Double-Blind, Placebo-Controlled Study to Evaluate the Efficacy and Safety of AT1001 for the Treatment of COVID-19 Related Multisystem Inflammatory Syndrome in Children (MIS-C)
Brief Title: AT1001 for the Treatment of COVID-19 Related MIS-C
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Decline in MISC cases
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Lael Yonker, M.D., Pulmonary Attending Physician, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2021P002143
Record Dates: First submitted 2021-08-09; First posted 2021-08-26 (Actual); Last update posted 2024-06-13 (Actual); Status verified 2024-06

CONDITIONS: Covid19; Multisystem Inflammatory Syndrome in Children
MeSH Terms: conditions — COVID-19; pediatric multisystem inflammatory disease, COVID-19 related | interventions — larazotide acetate

STUDY DESIGN:
Intervention Model Description: Placebo and drug arm (10 μg/kg/dose up to 500 μg/dose)
Who Masked: Participant, Investigator
Masking Description: Participant and investigator blinded, Pharmacy unblinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): Matching placebo will be administered orally four times a day (QID) to the standard of care for MIS-C.
  Interventions: Drug: Placebo
- Larazotide Acetate (Experimental): AT1001 10 μg/kg/dose up to 500 μg/dose (rounded to the nearest 50 μg) will be administered orally four times a day (QID) to the standard of care for MIS-C.
  Interventions: Drug: Larazotide Acetate

INTERVENTIONS:
Drug: Larazotide Acetate — AT1001 10 μg/kg/dose up to 500 μg/dose (rounded to the nearest 50 μg) will be administered orally four times a day (QID) to the standard of care for MIS-C.
  Other Names: AT1001
  Arms: Larazotide Acetate
Drug: Placebo — Matching placebo will be administered orally four times a day (QID) to the standard of care for MIS-C.
  Arms: Placebo

SUMMARY:
The primary aim of this study is to evaluate the efficacy and safety of AT1001 versus placebo in pediatric patients with SARS-CoV-2 infection who experience early signs of MIS-C and are at high risk of progression.

AT1001 10 μg/kg/dose up to 500 μg/dose (rounded to the nearest 50 μg) or matching placebo will be administered orally four times a day (QID) to the standard of care for MIS-C.

DETAILED DESCRIPTION:
This is a Phase 2a (Proof of Concept), randomized, double-blind, placebo-controlled study to evaluate the efficacy and safety of AT1001 for use in hospitalized pediatric patients diagnosed with MIS-C. Eligible participants (N=20) will be treated with AT1001 or matching placebo orally four times a day (QID) for up to 21 days as an add-on to standard of care.

The study includes three phases:

* Screening/Baseline: The main purpose of this phase is to determine if the participant meets entry criterion after obtaining informed consent and obtain baseline assessments.
* Treatment: Eligible participants will be treated with AT1001 or matching placebo 10 μg/kg/dose QID up to 500 μg/dose (rounded to the nearest 50 μg) for 21 days as an add-on to standard of care for MIS-C.
* Follow-up through 24 weeks: The participant will return for a follow-up visits during weekly clinic visits during Week 1 through Week 3, with monthly telemedicine visits at Week 4, Week 8, Week 16 and Week 20, and clinic visits at Week 12 and Week 24.

Safety monitoring, including physical examination, vitals, and clinical laboratory testing will be performed during the screening phase, periodically during treatment phase and at the follow-up phase. Adverse events and concomitant medications will be recorded during the entire study.

Total duration of the participants' participation in the study is approximately 24 weeks (with 21 days treatment period). Total duration of the study is projected to be 12 months, dependent on enrollment timeline.

ELIGIBILITY:
Inclusion Criteria:

1. Pediatric patients with or without comorbidity
2. Age ≥ 1 month to < 21 years
3. Confirmed MIS-C by signs and symptoms as detailed by the CDC Health Advisory (https://www.cdc.gov/mis-c/hcp/; May 14, 2020)

   1. Persistent fever/chills (>38.0°C for ≥24 hours, or report of subjective fever lasting ≥24 hours); AND
   2. One or more laboratory parameters (evidence of inflammation); AND,

   i) elevated C-reactive protein (CRP) ii) elevated erythrocyte sedimentation rate (ESR) iii) elevated ferritin iv) elevated lactic acid dehydrogenase (LDH) v) elevated d-dimer vi) elevated fibrinogen vii) elevated procalcitonin viii) elevated interleukin 6 (IL-6) ix) increased neutrophils x) reduced lymphocytes xi) low albumin c) Evidence of clinically severe illness requiring hospitalization, with multisystem (>2) organ involvement (cardiac, renal, respiratory, hematologic, gastrointestinal, dermatologic, or neurological)-MUST include GI symptoms, such as nausea, vomiting, diarrhea and/or abdominal pain; AND, d) No alternative plausible diagnoses; AND e) Positive for current or recent SARS-CoV-2 infection by RT-PCR, serology, or antigen test
4. Subject (or legal authorized representative) capable of understanding and signing an informed consent form and assent form, when appropriate.

Exclusion Criteria:

1. Female participants pregnant and/or lactating.
2. Female participant has childbearing potential and is unwilling to use an acceptable method of birth control for the duration of the study.
3. Participant has a significant co-morbid disease that by the Investigator's determination would make the participant unsuitable for enrollment, including unstable medical conditions.
4. Participation in any other clinical investigation using an experimental drug within 30 days prior to screening or intends to participate in another clinical study while participating in AT1001 MIS-C 101 study.
5. Have participated in a blood/plasma donation or blood loss greater than 400 mL within 90 days, or greater than 200 mL within 30 days prior to Screening.
6. Known hypersensitivity to any of the formulation components of AT1001.

Ages: 1 Month to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 12 (Actual)
Dates: Start 2021-10-01 (Actual); Primary Completion 2024-05-15 (Actual); Study Completion 2024-05-15 (Actual)

PRIMARY OUTCOMES:
Evaluate the efficacy and safety of AT1001 versus placebo on mitigating symptoms of MIS-C | 24 weeks
  • To evaluate the efficacy and safety of AT1001 versus placebo in pediatric patients with SARS-CoV-2 infection who experience early signs of MIS-C and are at high risk of progression.
Determine proportion of participants with improvement in MIS-C related GI symptoms and no progression of disease | 24 weeks
  Improvement in GI symptoms is defined as:
  * Improvement in PedsQL GI Symptoms Scales score ≥48 hours, as determined by patient or caregiver response.
  * AND improvement in clinical manifestation of GI symptoms, as documented by complete physical exam or clinical assessment and clinical laboratory tests or imaging.
  No Progression of MIS-C is defined as:
  * No involvement of additional organ involvement, as identified by clinical assessment and clinical laboratory tests or imaging.
  * AND no new onset of new or worsening GI symptoms for ≥48 hours including nausea, vomiting, diarrhea, loss of appetite, and/or abdominal pain, as determined by patient or caregiver symptom report or worsening PedsQL GI Symptoms Scales scores.

SECONDARY OUTCOMES:
Determine the impact of AT1001 on infectious and inflammatory markers of MIS-C | 24 weeks
  Secondary aims of this study include determining the impact of AT1001 on infectious and inflammatory markers of MIS-C.
Determine the impact of AT1001 on improvement in MIS-C symptoms for ≥48 hours, as determined by patient or caregiver symptom report on MIS-C Symptom Questionnaire. | 24 weeks
Determine the impact of AT1001 on length of stay in hospital (days from baseline to readiness to discharge). | 24 weeks
Determine the impact of AT1001 on re-presentation to medical care for MISC-related symptoms after discharge. | 24 weeks
Determine the impact of AT1001 on need for escalation of care (eg, transfer from hospital ward to ICU; supplemental oxygen; mechanical ventilation). | 24 weeks
  Transfer from hospital ward to ICU; supplemental oxygen; mechanical ventilation.
Determine the impact of AT1001 on change from baseline in additional organ system(s) involvement during acute presentation/hospitalization, as identified by clinical assessment and clinical laboratory tests. | 24 weeks
Determine the impact of AT1001 on change from baseline in levels of IgM, IgG, and IgA antibodies against SARS CoV-2. | 24 weeks
Determine the impact of AT1001 on change from baseline in levels of inflammatory markers (CRP, d-dimer, ferritin). | 24 weeks
Determine the impact of AT1001 on normalization of SARS-CoV-2 Spike, S1 and nucleocapsid. | 24 weeks
Determine the impact of AT1001 on change from baseline in levels of zonulin. | 24 weeks
Determine the impact of AT1001 on change in mortality (all causes) | 24 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No